CLINICAL TRIAL: NCT02026986
Title: Sleep Deprivation Reduces Tear Secretion and Impairs the Tear Film
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Young Joo Shin, MD, Hallym University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20131231
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: We Investigated the Effect of Sleep Deprivation on the Tear Film and Ocular Surface.

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sleep deprivation (Experimental): Ten subjects in the SD group were examined after a SD experiment in which they did not sleep for 24 h.
  Interventions: Behavioral: sleep deprivation
- control (No Intervention): The 10 subjects in the control group were not sleep deprived (had 8 h of sleep).

INTERVENTIONS:
Behavioral: sleep deprivation — sleep deprivation for one night
  Arms: sleep deprivation

SUMMARY:
Tear film consists of three layers including outer lipid layer, aqueous layer and inner mucin layer.1,2 Lipid layer protects the aqueous layer of tear film from evaporation and mucin layer adhere the tear film to ocular surface. Aqueous layer, which is produced in lacrimal glands, is the most important in the health of ocular surface. Reduction of aqueous tear secretion results in the disruption of homeostasis at ocular surface and leads to dry eye syndrome.2 Dry eye syndrome is a common ocular surface disease associated with symptoms of eye discomfort, grittness and visual disturbance.1,2 Dry eye syndrome disrupts normal homeostasis at the ocular surface resulting in epithelial damage, epithelial cell apoptosis, loss of goblet cells, and squamous metaplasia.1-3 The changes and inflammation of ocular surface subsequently lead to tear instability, which causes an increased tear osmolarity and aggravates the inflammatory cascades. This leads to a vicious cycle.2 The regulation of tear film secretion is under neural and hormonal control.4 Dry eye syndrome has been associated with diverse and multiple causes, including depressive disorder, drugs, hormonal status, and systemic diseases.2 Sleep deprivation (SD) is known to cause profound impair¬ments in executive function and vigilant attention.5,6 It is also reportedly associated with autonomic and endocrine functioning7-9 and has been shown to increase blood pressure and stress hormone levels and decrease parasympathetic tone.10,11 Tear secretion is regulated by neurological factors and hormones,12 and so SD may have an effect on the tear film and ocular surface. However, only a few studies have evaluated the effect of sleep on the tear film and ocular surface.

In this study, we investigated the effect of SD on the tear film and ocular surface.

DETAILED DESCRIPTION:
References

1. The definition and classification of dry eye disease: report of the Definition and Classification Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007;5:75-92.
2. Johnson ME, Murphy PJ. Changes in the tear film and ocular surface from dry eye syndrome. Prog Retin Eye Res. 2004;23:449-474.
3. Giacomo Savini, Pinita Prabhawasat, Takashi Kojima, Martin Grueterich, Edgar Espana, Eiki Goto. The challenge of dry eye diagnosis. Clin Ophthalmol. 2008; 2: 31-55.
4. Kamperis K, Hagstroem S, Radvanska E, Rittig S, Djurhuus JC. Excess diuresis and natriuresis during acute sleep deprivation in healthy adults. Am J Physiol Renal Physiol. 2010;299:F404-F411.
5. Mahler B, Kamperis K, Schroeder M, Frøkiær J, Djurhuus JC, Rittig S. Sleep deprivation induces excess diuresis and natriuresis in healthy children. Am J Physiol Renal Physiol. 2012;302:F236-F243.
6. McEwen BS. Sleep deprivation as a neurobiologic and physiologic stressor: Allostasis and allostatic load. Metabolism. 2006;55(10 Suppl 2):S20-S23.
7. Nascimento DC, Andersen ML, Hipólide DC, Nobrega JN, Tufik S. Pain hypersensitivity induced by paradoxical sleep deprivation is not due to altered binding to brain mu-opioid receptors. Behav Brain Res. 2007;178:216-220.
8. Everson CA. Functional consequences of sustained sleep deprivation in the rat. Behavioural Brain Research. 1995;69:43-54.
9. Kim JH, Kim JH, Nam WH, Yi K, Choi DG, Hyon JY, Wee WR, Shin YJ. Oral alcohol administration disturbs tear film and ocular surface. Ophthalmology. 2012;119:965-71.
10. Leproult R, Copinschi G, Buxton O, Van Cauter E. Sleep loss results in an elevation of cortisol levels the next evening. Sleep 1997;20:865-870.
11. Dartt DA. Neural regulation of lacrimal gland secretory processes: relevance in dry eye diseases. Prog Retin Eye Res. 2009;28:155-177.
12. The epidemiology of dry eye disease: report of the Epidemiology Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007;5:93-107.

ELIGIBILITY:
Inclusion Criteria:

* Twenty healthy young male volunteers aged 20-30 years

Exclusion Criteria:

* •Subjects with dry eye symptoms within the previous 6 months were excluded from the study.

  * Subjects have any systemic diseases such as systemic lupus, rheumatoid arthritis, Sjögren's syndrome or a history of ocular disease.
  * Subjects have disorder of lid margin, nasolacrimal duct, and cornea.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Tear osmolarity measurement | 1 day
  A microcapillary glass tube (Marienfeld, Lauda-Königshofen, Germany) was placed on the lower outer conjunctival sac. To avoid reflex tearing, the subjects were asked to direct their gaze supranasally. A total of 30 µL of tears was taken from the marginal tear strip. After centrifugation at 3000 rpm for 3 min, supernatants were obtained and the samples were stored at -80 degree. Tear osmolarity was measured using a Multi-OSMETTE 2430 (Precision Systems Inc., Natick, MA, USA).

SECONDARY OUTCOMES:
Visual analog pain score | 1 day
  Visual analog pain score Subjective discomfort or pain was graded numerically using the VAS. The scale range was 0 (absence of pain) to 10 (maximal pain). Subjects were asked to describe their symptoms using the VAS.
Tear break up time | 1 day
  Fluorescein was placed in the lower conjunctival sac using a fluorescein strip (HAAG-STREIT, Köniz, Switzerland), and the time between the last blink and the first appearance of a dark spot was measured using the cobalt blue light of a slit lamp. This procedure was repeated 3 times, and the average value was recorded.
Intraocular pressure | 1 day
  Intraocular pressure was measured by noncontact tonometer (CT-80, Topcon Corp., Tokyo, Japan). Intraocular pressure expressed in millimeters of mercury (mm Hg).
Schirmer's test | 1 day
  One drop of 0.5% proparacaine hydrochloride (Alcaine, Alcon, Forth Worth, TX, USA) was instilled in the conjunctival sac for topical anesthesia. In a silent room, filter paper (Color Bar, EagleVision, Memphis, TN, USA) was placed in the inferolateral one-third of the lower lid. Care was taken to prevent the paper from contacting the cornea. After 5 minutes, the level of strip wetting (in millimeters) was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Young Joo Shin, Principal Investigator — Hallym University
Locations (1):
- Hallym University, Kangnam Sacred Heart Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee YB, Koh JW, Hyon JY, Wee WR, Kim JJ, Shin YJ. Sleep deprivation reduces tear secretion and impairs the tear film. Invest Ophthalmol Vis Sci. 2014 May 15;55(6):3525-31. doi: 10.1167/iovs.14-13881. PMID 24833736